CLINICAL TRIAL: NCT02124577
Title: Development of Kinetic Biomarkers of Liver Fibrosis Based on Stable Isotope Mass Spectrometry Techniques for Measuring Nonalcoholic Fatty Liver Disease NAFLD)
Brief Title: Development of Kinetic Biomarkers of Liver Fibrosis Measuring NAFLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: KineMed (Industry)
Responsible Party: Principal Investigator, Rohit Loomba, Assistant Professor of Clinical Medicine, Division of Gastroenterology, Department of Medicine and, University of California, San Diego
Other Study IDs: 140338
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Biospecimen Retention: Samples With DNA — Stored specimen The specimens (serum, plasma, urine, stool, saliva, liver tissue, and DNA) collected as part of this study will be kept in Dr. Loomba' s locked research freezer at the Clinical Teaching Facility (CTF-building A).All collected data and patient charts will be maintained at the CTF building in a locked computer file with access available to the principal and study investigators only.
  All samples and data will be labeled with a code number. The name, address, social security number, date of birth and other personal identifiers will not be available on the sample, and we will not give out any information that identifies the patient to the researchers who use these samples and data.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a small preliminary study conducted to explore new methods for the potential of aiding in diagnosis of liver fibrotic disease as well as predicting disease progression. There will be a total of 4 visits spread out over approximately 8 weeks. You will be asked to drink "heavy water" during most of that time. "Heavy Water" also known as deuterated water, is physically and chemically very similar to ordinary drinking water. It tastes and feels exactly like regular water. It is odorless and has no known harmful effects at the doses given here. Heavy water occurs naturally, and is a minor component of the water we all ingest daily.

DETAILED DESCRIPTION:
Management of NASH and NAFLD remain a significant unmet medical challenge that is growing in importance as part of the obesity epidemic. Minimally invasive tools for monitoring disease progression and evaluating therapeutic interventions in NASH would be extremely valuable. Utilizing in vivo heavy water labeling, multiple pathways related to protein metabolism (fibrogenesis) and lipid metabolism can be quantified in human subjects. We have recently discovered that plasma lumicam synthesis represents a non-invasive kinetic biomarker of tissue fibrogenesis in patients with viral hepatitis. In addition, synthesis of fatty acids in plasma VLDL-triglycerides provide a window into hepatic lipid metabolism.

Stable isotopes have a long history as a safe, effective tracer for measuring synthesis of molecules in humans (1). Recently, new developments in stable isotope labeling techniques and advances in mass spectrometry have made in vivo kinetic measurement of slow metabolic processes possible. Through the use of 2H2O as the source of labeling, we and others have measured T-cell proliferation (2), mammary epithelial cell proliferation (3), prostate epithelial cell proliferation (4), triglyceride synthesis (5) and protein synthesis (6) in humans. We have recently evaluated this approach for the measurement of fibrogenesis patients with fibrotic liver disease.

Excess accumulation of collagen in the liver is termed fibrosis. Fibrosis is a common pathological feature of several chronic liver diseases (e.g. Hepatitis C, alcoholic liver disease, primary biliary sclerosis, drug/toxin induced liver disease, etc.). Currently, the standard method for detection of fibrosis is liver biopsy and histochemical analyses of tissue collagen content (8, 9). Although effective in diagnosing existing, advanced fibrosis, a single biopsy cannot measure current disease activity or predict rate of progression. To determine whether disease is progressing using current methods, a second biopsy is required. If significant additional collagen has accumulated since the first biopsy, this suggests that the disease is progressing. However, this measurement represents the history of the disease, not the current disease activity at the time of the second biopsy. There are also significant limitations in current methods, since changes in collagen pool size measurable by histochemistry cannot measure small changes in collagen content and intra-laboratory variability inherent in histochemical assays reduce their sensitivity (10, 11).

This stable isotope / mass spectrometry based method will be applied here for the quantification of fibrogenesis in vivo (from a bone marrow biopsy) and the identification of novel biomarkers of fibrogenesis in plasma in patients receiving investigational therapies.

If successful, this research will identify plasma proteins which can be easily measured by tandem mass spectrometry (LC/MS/MS) methods and whose synthesis rate reflects disease activity in the heart. Ideally, a set of markers related to NASH/ NAFLD will be developed that can detect and differentiate among multiple disease phenotypes, based on the kinetic signature measured in a single blood draw from a patient labeled with deuterated water.

The role of de novo lipogenesis (DNL) has been suggested by several clinical studies (Donnelly JCI 2005, Puri Hepatology 2009). DNL contributes significantly to the accumulation of lipid in NASH (Donnelly JCI 2005). Moreover DNL is elevated in many other inflammatory states and may be a useful marker of hepatic inflammation. DNL as well as hepatic TG assembly and cholesterogenesis are easily measured in plasma or dried blood spot samples from patients consuming 2H2O, after several days of labeling the plasma DNL reaches a steady state and reflects hepatic DNL rates.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18 years of age)
2. Adult male and female subjects, all races, ethnic groups, social and economic backgrounds and health status who are scheduled to undergo a liver biopsy as part of routine medical care will be included in the research.
3. Willingness to follow-up for 8 weeks
4. Written inform consent.

Exclusion Criteria:

1. Children younger than 18 will be excluded, since growth of liver tissue may confound measurements of collagen synthesis and cell proliferation due to normal turnover or disease.
2. The eligibility of patients will be determined by Dr. Rohit Loomba, MD or a referring physician at the time the potential subject is recommended to undergo a liver biopsy procedure as part of their medical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, age 18 or above, may have NAFLD or NASH-related cirrhosis or may serve as a control participant without this condition.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-05; Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
evaluate stable isotope/mass spectrometric methods | Baseline
  Our primary aim is to evaluate stable isotope/mass spectrometric methods for measuring in vivo liver collagen synthesis (fibrogenesis) and liver lipogenesis rates using liver biopsy specimens from patients with Non-Alcoholic Steatohepatitis (NASH)/ Nonalcoholic fatty liver disease (NAFLD).

SECONDARY OUTCOMES:
serum or urine markers of liver fibrogenesis that can be measured by the same stable isotope/mass spectrometric approach | Baseline
  Our secondary aim is to look for new serum or urine markers of liver fibrogenesis that can be measured by the same stable isotope/mass spectrometric approach in the same subjects. Subjects will drink the safe, non-toxic stable isotope heavy water (2H2O, deuterated water) prior to having a liver biopsy and providing urine and blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Loomba, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States